CLINICAL TRIAL: NCT07195695
Title: Beamion LUNG-3: A Randomized, Controlled, Multi-center Trial Evaluating Zongertinib as an Adjuvant Monotherapy Compared With Standard of Care in Patients With Early-stage, Resectable Non-small Cell Lung Cancer (Stage II-IIIB) Harboring Tyrosine Kinase Domain Activating HER2 Mutations
Brief Title: Beamion LUNG-3: A Study to Test Whether Zongertinib Helps People With Surgically Removed, Non-small Cell Lung Cancer With HER2 Mutations Compared With Standard Treatment
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1479-0032; U1111-1320-6149 (Registry Identifier: WHO - International Clinical Trials Registry Platform (ICTRP)); 2025-521284-12-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-25; First posted 2025-09-29 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; atezolizumab; durvalumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Zongertinib treatment arm (Experimental)
  Interventions: Drug: Zongertinib
- Standard of Care (SoC) treatment arm (Active Comparator)
  Interventions: Drug: Pembrolizumab; Drug: Atezolizumab; Drug: Durvalumab; Drug: Nivolumab

INTERVENTIONS:
Drug: Zongertinib — Zongertinib
  Other Names: BI 1810631, Hernexeos®
  Arms: Zongertinib treatment arm
Drug: Pembrolizumab — Pembrolizumab
  Arms: Standard of Care (SoC) treatment arm
Drug: Atezolizumab — Atezolizumab
  Arms: Standard of Care (SoC) treatment arm
Drug: Durvalumab — Durvalumab
  Arms: Standard of Care (SoC) treatment arm
Drug: Nivolumab — Nivolumab
  Arms: Standard of Care (SoC) treatment arm

SUMMARY:
This study is open to adults 18 years and older who have early-stage non-small cell lung cancer (NSCLC). Their cancer must have a specific change in a gene called HER2. Genes provide the instructions for making proteins, and this change leads to a faulty HER2 protein. People can join if their lung cancer was removed by surgery, and they have already received certain other anti-cancer treatments. The purpose of this study is to find out if a study medicine called zongertinib helps people with this type of cancer live longer without their cancer coming back after surgery, when compared to standard treatment. Zongertinib is being developed to target the faulty HER2 protein, which can cause cancer cells to grow.

In this study, participants are assigned by chance to one of two treatment groups, with an equal chance of being in either group. One group takes the study medicine, zongertinib, by mouth once a day for up to 3 years. The other group receives a standard treatment, chosen by their doctor. This standard treatment may be an immunotherapy medicine given by infusion into a vein every 3 or 4 weeks for up to 1 year, or regular check-ups without active study medicine (observation).

Participants can be in this study for up to about 11 years. During this time, they visit the study site regularly for check-ups and study-related tests. The frequency of these visits varies depending on their treatment and how long they have been in the study. In addition to visits at the study site, participants in some treatment groups will also have phone calls with the study team every 3 weeks to check on their health between their scheduled visits.

Doctors check for any signs of cancer coming back using imaging scans (like CT or MRI scans); these scans are generally done every 3 months for the first 2 years, then every 6 months for the next 3 years, and then yearly. Participants also fill in questionnaires about their overall wellbeing, health and symptoms. Throughout the study, doctors also check participants' health and note any unwanted effects.

ELIGIBILITY:
Inclusion criteria:

1. Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial
2. Patients must be ≥18 years old or over the legal age of consent in their country
3. Male or female patients. Women of childbearing potential (WOCBP) must be ready and able to use dual highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in the patient information and in the study protocol
4. HER2 mutation: Documented Tyrosine kinase domain (TKD) activating Human epidermal growth factor receptor 2 (HER2) mutations
5. Histology and tumor sample: Histologically confirmed diagnosis of primary NSCLC
6. An archival tumor tissue sample must be submitted to the central laboratory after inclusion of the patient to retrospectively confirm the HER2 status
7. Staging: Pretherapeutic classification not exceeding Stage IIIB
8. Performance status and organ function:

   * Eastern Cooperative Oncology Group (ECOG) score of 0 or 1
   * Adequate organ function based on laboratory values Further inclusion criteria apply.

Exclusion criteria:

1. Diagnosis of NSCLC with mixed histology/positive neuroendocrine markers (synaptophysin/CD56)
2. Major surgery (major according to the investigator's assessment) performed within 4 weeks prior to randomization
3. Treatment with radiation therapy for primary NSCLC
4. Co-occurring actionable mutation with approved targeted therapy (e.g. Epidermal growth factor receptor (EGFR) or Anaplastic lymphoma kinase (ALK))
5. Any investigational drug within 5 half-lives of the compound or any of its related material, if known
6. History or presence of

   * Active or known pre-existing or history of non-infectious interstitial lung disease/pneumonitis
   * Active infectious disease requiring systemic therapy
   * Uncontrolled gastrointestinal disorders affecting drug intake/absorption
   * Previous or concomitant malignancies within the last 3 years, except certain effectively treated cancers
   * Significant and/or uncontrolled cardiovascular abnormalities, QT interval corrected for heart rate by Fridericia formula (QTcF) >470 msec, or ejection fraction <50% Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2026-01-16 (Actual); Primary Completion 2032-02-26 (Estimated); Study Completion 2036-09-02 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) by investigator's assessment | up to 8 years and 5 months
  DFS is defined as the time from randomization until recurrence of tumor or death from any cause, whichever occurs earlier

SECONDARY OUTCOMES:
Key secondary endpoint: Overall survival (OS), defined as the time from randomization until death from any cause | up to 8 years and 5 months
Occurrence of trial-related Adverse Events (AEs) ≥ Grade 3 from first treatment administration (or from randomization for patients in the observation arm) until the earliest of tumor recurrence or 3 years since treatment start | up to 3 years
  AEs are graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0

CONTACTS AND LOCATIONS:
Locations (184):
- United States (23):
  - ClinRé 001-022 (Premier Cancer Care and Infusion Center), Fresno, California
  - OPN Healthcare, Inc., Glendale, California
  - Sutter Health, Roseville, California
  - Sarcoma Oncology Center, Santa Monica, California
  - University of California Los Angeles, Santa Monica, California
  - Northern California Kaiser Permanente, Vallejo, California
  - George Washington University Cancer Center, Washington D.C., District of Columbia
  - Mid Florida Hematology and Oncology Center, Orange City, Florida
  - Piedmont Cancer Institute, Atlanta, Georgia
  - Northwest Georgia Oncology Centers, Marietta, Georgia
  - Saint Alphonsus Regional Medical Center - Boise, Boise, Idaho
  - Northwestern University, Chicago, Illinois
  - University of Illinois Hospital and Health Sciences System, Chicago, Illinois
  - Duly Health and Care - Lisle, Lisle, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Cancer Care Specialists, Reno, Nevada
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Laura & Isaac Perlmutter Cancer Center at NYU Langone Health, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Providence Cancer Institute, Portland, Oregon
  - Hendrick Health, Abilene, Texas
  - Community Cancer Trials of Utah, Ogden, Utah
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
- Argentina (5):
  - Centro de Investigaciones Médicas y Desarrollo LC S.R.L. (LC Investigación), CABA
  - Hospital Britanico de Buenos Aires, CABA
  - Centro Oncologico Korben, CABA
  - Clinica Adventista Belgrano, CABA
  - Instituto Medico Especializado Alexander Fleming, Capital Federal
- St John of God Subiaco Hospital, Subiaco, Western Australia, Australia
- Austria (2):
  - Medical University of Innsbruck, Innsbruck
  - Clinic Floridsdorf, Vienna
- Belgium (3):
  - Edegem - UNIV UZ Antwerpen, Edegem
  - UZ Leuven, Leuven
  - Centre Hospitalier Universitaire de Liège, Liège
- Brazil (7):
  - Hospital de Amor, Barretos
  - NewData Clinical Research - Maceió, Maceió
  - Centro de Pesquisa Oncology Natal, Natal
  - Centro Gaúcho Integrado de Oncologia, Hematologia, Ensino e Pesquisa, Porto Alegre
  - CEPHO - Centro de Estudos e Pesquisas em Hematologia e Oncologia, Santo André
  - ICESP - Instituto do Cancer do Estado de Sao Paulo, São Paulo
  - A.C. Camargo, São Paulo
- Canada (2):
  - Cross Cancer Institute (University of Alberta), Edmonton, Alberta
  - Princess Margaret Cancer Centre, Toronto, Ontario
- Chile (2):
  - Centro de Estudios Clinicos SAGA, Providencia
  - Bradford Hill- Centro de Investigación Clínica, Recoleta
- China (28):
  - China-Japan Friendship Hospital, Beijing
  - Beijing Chest Hospital, Capital Medical University, Beijing
  - The First Hospital of Jilin University, Changchun
  - Xiangya Hospital, Central South University, Changsha
  - Hunan Province Tumor Hospital, Changsha
  - Sichuan Cancer Hospital, Chengdu
  - West China Hospital, Sichuan University, Chengdu
  - The First Affiliated Hospital,Sun Yat-sen University, Guangzhou
  - The First Affiliated Hospital, Zhejiang University, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Shandong Cancer Hospital, Jinan
  - Yunnan Provincial Tumor Hospital, Kunming
  - Linyi Cancer Hospital, Linyi
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Nanjing Drum Tower Hospital, Nanjing
  - Ningbo Second Hospital, Ningbo
  - Shanghai East Hospital, Shanghai
  - Shanghai Pulmonary Hospital, Shanghai
  - Hebei Provincial Tumor Hospital, Shijiazhuang
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Taizhou Hospital of Zhejiang Province, Taizhou
  - Tianjin Cancer Hospital, Tianjin
  - Tianjin Medical University General Hospital, Tianjin
  - Wuhan Union Hospital, Wuhan
  - Affiliated Hospital, Xuzhou Medical college, Xuzhou
  - Northern Jiangsu People's Hospital, Yangzhou
  - Henan Cancer Hospital, Zhengzhou
- Sjællands Universitetshospital, Roskilde, Denmark
- Egypt (2):
  - National Cancer Institute, Cairo University, Cairo
  - Shefaa El Orman Oncology Hospital, Luxor
- France (6):
  - HOP Louis Pradel, Bron
  - HOP Nord Laennec, Nantes
  - HOP Pontchaillou, Rennes
  - Centre Régional de Lutte Contre le Cancer Paul Stauss, Strasbourg
  - Hôpital Larrey - CHU de Toulouse, Toulouse
  - INS Gustave Roussy, Villejuif
- Germany (8):
  - Universitätsklinikum Köln (AöR), Cologne
  - Klinikum Esslingen, Esslingen am Neckar
  - Varisano LungenZentrum (VLZ), Frankfurt
  - Asklepios Fachkliniken München-Gauting, Gauting
  - LungenClinic Grosshansdorf GmbH, Großhansdorf
  - Thoraxklinik-Heidelberg gGmbH am Universitätsklinikum Heidelberg, Heidelberg
  - Pius-Hospital, Oldenburg, Oldenburg
  - Universitätsklinikum Würzburg AÖR, Würzburg
- Greece (3):
  - Henry Dunant Hospital, Athens, Athens
  - Chest Hospital of Athens "Sotiria", Athens
  - University General Hospital Attikon, Athens
- Hong Kong (4):
  - Queen Elizabeth Hospital-Hong Kong-51727, Hong Kong
  - Prince of Wales Hospital-Hong Kong-20715, Hong Kong
  - Princess Margaret Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
- Israel (5):
  - Rambam Health Care Campus, Haifa
  - Shaare Zedek Medical Center, Jerusalem 91031, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Sheba Medical Center, Ramat Gan
  - Sourasky Medical Center, Tel Aviv
- Italy (8):
  - Istituto Tumori Giovanni Paolo II, Bari
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Humanitas Istituto Clinico Catanese S.p.A., Misterbianco (CT)
  - Istituto Nazionale IRCCS Tumori Fondazione Pascale, Napoli
  - AOU San Luigi Gonzaga, Orbassano (TO)
  - Istituti Fisioterapici Ospitalieri, Roma
  - Istituto Clinico Humanitas, Rozzano (MI)
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona
- Japan (25):
  - Aichi Cancer Center Hospital, Aichi, Nagoya
  - Fujita Health University Hospital, Aichi, Toyoake
  - National Cancer Center Hospital East, Chiba, Kashiwa
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Hospital of the University of Occupational and Environmental Health, Fukuoka, Kitakyushu
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - Hokkaido Cancer Center, Hokkaido, Sapporo
  - Kitasato University Hospital, Kanagawa, Sagamihara
  - Kanagawa Cancer Center, Kanagawa, Yokohama
  - Sendai Kousei Hospital, Miyagi, Sendai
  - Niigata Cancer Center Hospital, Niigata, Niigata
  - Okayama University Hospital, Okayama, Okayama
  - Kansai Medical University Hospital, Osaka, Hirakata
  - Osaka International Cancer Institute, Osaka, Osaka
  - Kindai University Hospital, Osaka, Sakai
  - National Hospital Organization Kinki-Chuo Chest Medical Center, Osaka, Sakai
  - Saitama Medical University International Medical Center, Saitama, Hidaka
  - Saitama Cancer Center, Saitama, Kitaadachi-gun
  - Shizuoka Cancer Center, Shizuoka, Sunto-gun
  - Jichi Medical University Hospital, Tochigi, Shimotsuke
  - Juntendo University Hospital, Tokyo, Bunkyo-ku
  - National Cancer Center Hospital, Tokyo, Chuo-ku
  - Japanese Foundation for Cancer Research, Tokyo, Koto-ku
  - Tokyo Medical University Hospital, Tokyo, Shinjuku-ku
  - Wakayama Medical University Hospital, Wakayama, Wakayama
- Mexico (4):
  - Centro Oncologico Internacional, Jalisco
  - Centro de Infusion Profesional Integral (CIPI), Mexico City
  - Instituto Nacional de Cancerologia, México
  - Centro Medico Zambrano Hellion, Monterrey
- Nederlands Kanker Instituut - Antoni van Leeuwenhoek Amsterdam (METC AVL), Amsterdam, Netherlands
- Portugal (4):
  - Hospital CUF Tejo, Lisbon
  - Hospital da Luz, Lisbon
  - Hospital CUF Porto, Porto
  - IPO Porto Francisco Gentil, EPE, Porto
- Romania (4):
  - Lotus Med, Bucharest
  - Memorial Healthcare International, Bucharest
  - Ovidius Clinical Hospital S.R.L, Ovidiu
  - Polaris Medical S.A., Suceagu/ Cluj Napoca
- South Korea (8):
  - National Cancer Center, Goyang
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, St.Vincent's Hospital, Suwon
  - Ajou University Hospital, Suwon
- Spain (14):
  - Hospital del Mar, Barcelona
  - Hospital Universitari Vall D Hebron, Barcelona
  - Hospital Universitario De Burgos, Burgos
  - Hospital General Universitario de Elche, Elche
  - Hospital Jerez de la Frontera, Jerez de la Frontera
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Puerta de Hierro, Majadahonda
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Complejo Hospitalario de Navarra, Pamplona
  - Salut Sant Joan de Reus, Reus
  - Hospital Virgen del Rocío, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
- Sweden (2):
  - Sahlgrenska Universitetsjukhuset, Gothenburg
  - Karolinska Universitetssjukhuset Solna, Stockholm
- Taiwan (6):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan
- Sağlık Bilimleri Üniversitesi Gülhane Eğitim ve Araştırma Hastanesi, Ankara, Turkey (Türkiye)
- United Kingdom (5):
  - Western General Hospital, Edinburgh
  - Guy's Hospital, London
  - The Royal Marsden Hospital, Chelsea, London
  - The Christie, Manchester
  - The Royal Marsden Hospital, Sutton, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents - upon signing of a "Document Sharing Agreement". For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.clinicalstudies.boehringer-ingelheim.com/msw/datatransparency